CLINICAL TRIAL: NCT00605111
Title: Efficacy and Safety of Initiation of Biphasic Insulin Aspart 30 Treatment in Subjects With Type 2 Diabetes Mellitus Failing OAD Therapy
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3021
Record Dates: First submitted 2008-01-18; First posted 2008-01-30 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the efficacy and safety of biphasic insulin aspart 30 as start insulin in subjects with type 2 diabetes failing OAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 24 months
* BMI between 18 and 30 kg/m2
* Insulin naive subjects
* OAD treatment with max two OADs alone or combined with other therapy
* HbA1c between 7-12%

Exclusion Criteria:

* Type 1 diabetes
* Receipt of any investigational drug within the last three months prior to this trial
* Current or previous treatment with thiazolidiones within the last 6 months
* OAD treatment with three or more OADs within the last 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2003-12; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 11 weeks of treatment

SECONDARY OUTCOMES:
The proportion of subjects achieving treatment target of HbA1c below 7% | at 11 and 24 weeks
8-point plasma glucose profiles | performed at 11 and 24 weeks
FPG | at 11 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- Australia (5):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Fitzroy
  - Novo Nordisk Investigational Site, Garran
  - Novo Nordisk Investigational Site, Stones Corner
- Hong Kong (2):
  - Novo Nordisk Investigational Site, Hong Kong Island
  - Novo Nordisk Investigational Site, Shatin, New Territories
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Georgetown, Penang
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
- Philippines (2):
  - Novo Nordisk Investigational Site, Cebu City
  - Novo Nordisk Investigational Site, Quezon City
- Novo Nordisk Investigational Site, Singapore, Singapore
- Taiwan (2):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Kaoshiung
- Novo Nordisk Investigational Site, Bangkok, Thailand

REFERENCES:
- [Result] Bebakar WM, Chow CC, Kadir KA, Suwanwalaikorn S, Vaz JA, Bech OM; BIAsp-3021 study group. Adding biphasic insulin aspart 30 once or twice daily is more efficacious than optimizing oral antidiabetic treatment in patients with type 2 diabetes. Diabetes Obes Metab. 2007 Sep;9(5):724-32. doi: 10.1111/j.1463-1326.2007.00743.x. Epub 2007 Jun 26. PMID 17593237
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com